CLINICAL TRIAL: NCT05705427
Title: Simplifying Hepatitis B Care in Pregnancy by Combining Birth-dose Vaccine and Tenofovir: The COMBAT HBV Feasibility Trial
Brief Title: The COMBAT HBV Feasibility Trial
Acronym: COMBAT-HBV
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Doris Duke Charitable Foundation (Other); Université Protestant au Congo (Unknown); Abbott (Industry); Albert Einstein College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 22-1492
Record Dates: First submitted 2023-01-20; First posted 2023-01-30 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Hepatitis B; Vertical Transmission of Infectious Disease
Keywords: Prevention of mother-to-child transmission; Hepatitis B birth-dose vaccine; Tenofovir disoproxil fumarate
MeSH Terms: conditions — Hepatitis B | interventions — Tenofovir; Engerix-B

STUDY DESIGN:
Intervention Model Description: Pregnant women will be randomized at the time of enrollment (at 28-32 weeks' gestation) in a 1:1 ratio to receive tenofovir disoproxil fumarate (TDF) vs placebo, with an expected 140 women in the TDF arm and 140 in the placebo arm. A permuted block randomization technique will be employed to ensure equal distribution between the two arms at the two maternity centers. A biostatistician from the University of North Carolina (UNC) will design the randomization scheme, which will utilize the randomization-and-concealment feature within the REDCap database; the biostatistician will not be directly involved in study enrollment activities. REDCap personnel at UNC will ensure proper design and use of the randomization-and-concealment feature, and study personnel will receive training on the randomization process prior to study roll-out.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The trial will be double-blinded, with study staff and participants blinded to allocation to the TDF vs placebo arm. Blinding to medication type will be achieved via use of over-encapsulation of TDF and placebo pills. Laboratory technicians who perform point-of-care hepatitis B core related antigen testing, HBV viral load testing and hepatitis B e antigen testing will be blinded to study arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tenofovir disoproxil fumarate (TDF) arm (Experimental): 140 pregnant women in the experimental arm will receive tenofovir disoproxil fumarate (TDF) 300 milligrams (mg) daily, beginning at 28-32 weeks' gestation and continuing through 4 weeks' postpartum. Infants born to these women will be included in this arm and will receive a birth-dose of hepatitis B vaccine.
  Interventions: Drug: Tenofovir Disoproxil Fumarate 300 MG; Biological: Hepatitis B monovalent vaccine
- Placebo arm (Placebo Comparator): 140 pregnant women in the placebo arm will receive a placebo pill daily, beginning at 28-32 weeks' gestation and continuing through 4 weeks' postpartum. Infants born to these women will be included in this arm and will receive a birth-dose of hepatitis B vaccine.
  Interventions: Biological: Hepatitis B monovalent vaccine; Drug: Placebo

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate 300 MG — Pregnant women in the experimental arm will receive TDF daily beginning in the 3rd trimester of pregnancy and continuing through 1 month postpartum.
  Other Names: Viread
  Arms: Tenofovir disoproxil fumarate (TDF) arm
Biological: Hepatitis B monovalent vaccine — All infants born to women in the study will receive a birth-dose hepatitis B vaccine.
  Other Names: Hepatitis B birth-dose vaccine; Engerix-B
Drug: Placebo — Pregnant women in the placebo arm will receive a placebo pill daily beginning in the 3rd trimester of pregnancy and continuing through 1 month postpartum.
  Arms: Placebo arm

SUMMARY:
This is a double-blind, randomized placebo-controlled trial (RCT) of a prophylaxis-for-all approach to prevention of mother-to-child transmission (PMTCT) of hepatitis B virus (HBV) in the Democratic Republic of Congo (DRC). HBV-infected pregnant women will be randomized to either receive tenofovir or placebo beginning at 28-32 weeks' gestation and continuing through 4 weeks' postpartum. Women will be followed every 4-6 weeks throughout the prenatal and postpartum period to evaluate for side effects related to the medication. Infants will receive a birth-dose of HBV vaccine, ideally within 24 hours. Participants will be followed longitudinally through 6 months' postpartum.

DETAILED DESCRIPTION:
The overall study design is a randomized, double-blind, placebo-controlled trial among two groups of mother-infant dyads: women who receive TDF vs placebo in late pregnancy and the postpartum period (beginning at 28-32 weeks' gestation and continuing through 4 weeks' postpartum). While official World Health Organization (WHO) recommendations are to continue TDF at least through delivery, a range from delivery through 12 weeks' postpartum is possible; the investigators will continue therapy through 4 weeks' postpartum in this study. This feasibility trial will evaluate the acceptability, safety and preliminary effectiveness of a TDF-for-all approach to prevent MTCT of HBV in low-resource settings. HBsAg-positive pregnant women will be enrolled at 28-32 weeks' gestation, and will present for regular medication checks, with a study closeout visit at 24 weeks' postpartum. Study activities at monthly medication checks will include medication refills, assessment of adherence (via pill counts and verbal surveys), and evaluation for side effects. All infants will receive a birth-dose of HBV vaccine within 24 hours of life. MTCT of HBV will be defined as the proportion of infants with positive HBsAg testing at 6 months. This pilot study will provide preliminary data for sample size calculations, including safety and effectiveness data, to prepare for larger RCTs to determine the effectiveness of a tenofovir-for-all approach, as well as the added benefit of tenofovir over birth-dose vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women ≥18 years of age who present for routine prenatal care between 28-32 weeks' gestation and who test HBV-positive by point-of-care hepatitis B surface antigen test. Women must intend to seek maternity and postpartum care exclusively at one of the Kinshasa-based study maternity centers.
* Infants born to enrolled women will be included in the study

Exclusion Criteria:

* Individuals with abnormal creatinine by point-of-care testing
* Any woman who plans to move outside of Kinshasa Province during the study period.
* Any HIV-positive individual, determined by routine point-of-care screening at antenatal care visits

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2023-08-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Safety (Pregnant Women): Number of Pregnant Women With Adverse Effects Related to Study Medications | Up to study close-out visit, or up to 12 months
  Safety of TDF prophylaxis in pregnant women, defined as a composite of adverse events (# mild adverse events [AEs], # moderate-to-severe AEs), presence of side effects and alanine aminotransferase elevations ≥ 5x upper limit of normal
Safety (Infants): Number of Infants with Adverse Effects Related to Study Medications | At delivery
  Safety of maternal TDF for infants, defined as a composite of: Birth weight (grams), mid-upper arm circumference (centimeters), gestational age at delivery (weeks and days), delivery mode (vaginal vs C-section), APGAR scores (0-10), # of adverse events
Feasibility (Recruitment): Number of Eligible Participants Who Were Enrolled in the Study | Up to study close-out visit, or up to 12 months
  Recruitment is indicative of the number of pregnant women who are screened versus those actually enrolled in the study.
Feasibility (Refusal): Number of Eligible Participants Who Refused to Enroll in the Study | Up to study close-out visit, or up to 12 months
  Refusal will be defined as the number of individuals who refuse enrollment upon initial recruitment.
Feasibility (Withdrawal): Number of Enrolled Participants Who Withdraw from the Study | Up to study close-out visit, or up to 12 months
  Withdrawal is indicative of the number of enrolled participants who choose not to continue study activities after having been enrolled.
Feasibility (Retention): Number of Enrolled Participants Who Remain in the Study Through 6 Months Postpartum | Up to study close-out visit, or up to 12 months
  Retention is defined as the number of participants who remain in the study through the 6-month postpartum visit.
Feasibility (Maintenance): Proportion of Study Visits Completed Per Participant | Up to study close-out visit (12 months)
  Adherence to study visits and procedures, defined as proportion of the actual number of visits attended divided by the expected study visits (8) and multiplied by 100.
Acceptability (Lab Testing): Number of Mothers With Lab Testing Acceptability Scores >80% | Upon study close-out visit, or up to 12 months
  Number of mothers who report the process of undergoing lab draws as "acceptable" in the exit survey. Range 0-100%, with 0% being unacceptable and 100% being acceptable.
Acceptability (Medication): Number of Mothers With Medication Acceptability Scores >80% | Upon study close-out visit, or up to 12 months
  Number of mothers who report the process of taking the study medication as "acceptable" in the exit survey. Range 0-100%, with 0% being unacceptable and 100% being acceptable.
Preliminary Effectiveness: Number of Infants With HBV Positivity by Rapid Diagnostic Testing at 6 Months of Life to Indicate Mother-to-Child Transmission of HBV | Measured at 6 months after birth
  Mother-to-child transmission of HBV is defined as HBsAg positivity in the infant at 6 months of life.

SECONDARY OUTCOMES:
Sensitivity of the Hepatitis B Core-Related Antigen Test | Measured at Enrollment
  Sensitivity will be defined as the number of true positive tests divided by the sum of the true positives and false negatives.
Specificity of the Hepatitis B Core-Related Antigen Test | Measured at Enrollment
  Specificity will be defined as the number of true negative tests divided by the sum of the true negatives and the false positives.

CONTACTS AND LOCATIONS:
Overall Officials: Peyton Thompson, MD, MSCR, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Université Protestant au Congo, Kinshasa, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: Yes
Datasets will not be made publicly available because they contain protected health information. However, the authors will share de-identified participant data, alongside the study protocol, statistical analysis plan, and analytic code, upon reasonable request and with approval by an independent review committee (ie, learned intermediary). An executed Data Use/Sharing agreement with the University of North Carolina at Chapel Hill (UNC-CH) is required before data will be shared
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available from 9 to 36 months after publication.
Access Criteria: Interested individuals can request de-identified data with approval from an independent review committee, which will be shared upon execution of a Data Use/Sharing Agreement with UNC-CH.